CLINICAL TRIAL: NCT02559206
Title: A Phase 2b, Randomized, Double-blind, Double-dummy, Placebo-controlled, Parallel-group, Dose-range-finding Study of Two Delayed Release Formulations of Linaclotide Administered Orally for 12 Weeks to Patients With Irritable Bowel Syndrome With Constipation
Brief Title: Trial of Linaclotide in Patients With Irritable Bowel Syndrome With Constipation (IBS-C)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ironwood Pharmaceuticals, Inc. (Industry)
Collaborators: Forest Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MCP-103-204
Record Dates: First submitted 2015-09-22; First posted 2015-09-24 (Estimated); Results first posted 2020-04-24 (Actual); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Irritable Bowel Syndrome With Constipation
MeSH Terms: interventions — linaclotide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (8):
- 30 μg linaclotide DR1 and placebo (Experimental)
  Interventions: Drug: Linaclotide
- 100 μg linaclotide DR1 and placebo (Experimental)
  Interventions: Drug: Linaclotide
- 300 μg linaclotide DR1 and placebo (Experimental)
  Interventions: Drug: Linaclotide
- 30 μg linaclotide DR2 and placebo (Experimental)
  Interventions: Drug: Linaclotide
- 100 μg linaclotide DR2 and placebo (Experimental)
  Interventions: Drug: Linaclotide
- 300 μg linaclotide DR2 and placebo (Experimental)
  Interventions: Drug: Linaclotide
- 290 μg linaclotide IR and placebo (Experimental)
  Interventions: Drug: Linaclotide
- Placebo (Placebo Comparator)
  Interventions: Drug: Matching Placebo

INTERVENTIONS:
Drug: Linaclotide — Oral, once daily
  Arms: 100 μg linaclotide DR1 and placebo; 100 μg linaclotide DR2 and placebo; 290 μg linaclotide IR and placebo; 30 μg linaclotide DR1 and placebo; 30 μg linaclotide DR2 and placebo; 300 μg linaclotide DR1 and placebo; 300 μg linaclotide DR2 and placebo
Drug: Matching Placebo — Oral, once daily
  Arms: Placebo

SUMMARY:
The objectives of this study are to evaluate the safety, efficacy, and dose response of two delayed release formulations of linaclotide (DR; DR formulation 1 is DR1; DR formulation 2 is DR2) administered orally to patients with irritable bowel syndrome with constipation (IBS-C). Additional objectives include understanding how the two DR formulations compare with each other and with the FDA-approved 290 μg LINZESS® (the immediate release [IR] formulation of linaclotide).

ELIGIBILITY:
Inclusion Criteria:

* Patient has completed a colonoscopy according to the American Gastroenterological Association (AGA) criteria, with no clinically significant findings
* Patient has no clinically significant findings on a physical examination and clinical laboratory tests
* Patient meets protocol criteria for diagnosis of IBS-C
* Patient demonstrates continued IBS-C through Pretreatment Period
* Patient maintains a minimum level of compliance with daily diary

Exclusion Criteria:

* Patient has history of loose or watery stools
* Patient has symptoms of or been diagnosed with a medical condition that may contribute to abdominal pain
* Patient has a structural abnormality of the gastrointestinal (GI) tract or a disease or condition that can affect GI motility
* Patient has any protocol-excluded or clinically significant medical or surgical history that could confound the study assessments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 759 (Actual)
Dates: Start 2015-10-22 (Actual); Primary Completion 2016-09-30 (Actual); Study Completion 2016-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Chamberlin, MD, Study Chair — Ironwood Pharmaceuticals, Inc.
Locations (64):
- United States (64):
  - Ironwood Investigational Site, Huntsville, Alabama
  - Ironwood Investigational Site, Phoenix, Arizona
  - Ironwood Investigational Site, Tucson, Arizona
  - Ironwood Investigational Site, North Little Rock, Arkansas
  - Ironwood Investigational Site, Anaheim, California
  - Ironwood Investigational Site, Chula Vista, California
  - Ironwood Investigational Site, Garden Grove, California
  - Ironwood Investigational Site, La Mesa, California
  - Ironwood Investigational Site, Newport Beach, California
  - Ironwood Investigational Site, Orange, California
  - Ironwood Investigational Site, San Diego, California
  - Ironwood Investigational Site, Thousand Oaks, California
  - Ironwood Investigational Site, Colorado Springs, Colorado
  - Ironwood Investigational Site, Bristol, Connecticut
  - Ironwood Investigational Site, Waterbury, Connecticut
  - Ironwood Investigational Site, Hialeah, Florida
  - Ironwood Investigational Site, Kissimmee, Florida
  - Ironwood Investigational Site, Miami, Florida
  - Ironwood Investigational Site, Orlando, Florida
  - Ironwood Investigational Site, South Miami, Florida
  - Ironwood Investigational Site, Tampa, Florida
  - Ironwood Investigational Site, West Palm Beach, Florida
  - Ironwood Investigational Site, Atlanta, Georgia
  - Ironwood Investigational Site, Oakwood, Georgia
  - Ironwood Investigational Site, Sandy Springs, Georgia
  - Ironwood Investigational Site, Evansville, Indiana
  - Ironwood Investigational Site, Bastrop, Louisiana
  - Ironwood Investigational Site, Metairie, Louisiana
  - Ironwood Investigational Site, Shreveport, Louisiana
  - Ironwood Investigational Site, Baltimore, Maryland
  - Ironwood Investigational Site, Chevy Chase, Maryland
  - Ironwood Investigational Site, Boston, Massachusetts
  - Ironwood Investigational Site, Watertown, Massachusetts
  - Ironwood Investigational Site, Chesterfield, Michigan
  - Ironwood Investigational Site, Wyoming, Michigan
  - Ironwood Investigational Site, Jackson, Mississippi
  - Ironwood Investigational Site, St Louis, Missouri
  - Ironwood Investigational Site, Bozeman, Montana
  - Ironwood Investigational Site, Las Vegas, Nevada
  - Ironwood Investigational Site, Brooklyn, New York
  - Ironwood Investigational Site, Charlotte, North Carolina
  - Ironwood Investigational Site, Concord, North Carolina
  - Ironwood Investigational Site, Davidson, North Carolina
  - Ironwood Investigational Site, Fayetteville, North Carolina
  - Ironwood Investigational Site, Wilmington, North Carolina
  - Ironwood Investigational Site, Winston-Salem, North Carolina
  - Ironwood Investigational Site, Cincinnati, Ohio
  - Ironwood Investigational Site, Mentor, Ohio
  - Ironwood Investigational Site, Xenia, Ohio
  - Ironwood Investigational Site, Pittsburgh, Pennsylvania
  - Ironwood Investigational Site, Dakota Dunes, South Dakota
  - Ironwood Investigational Site, Bristol, Tennessee
  - Ironwood Investigational Site, Chattanooga, Tennessee
  - Ironwood Investigational Site, Knoxville, Tennessee
  - Ironwood Investigational Site, Arlington, Texas
  - Ironwood Investigational Site, Beaumont, Texas
  - Ironwood Investigational Site, El Paso, Texas
  - Ironwood Investigational Site, Houston, Texas
  - Ironwood Investigational Site, San Antonio, Texas
  - Ironwood Investigational Site, Ogden, Utah
  - Ironwood Investigational Site, Sandy City, Utah
  - Ironwood Investigational Site, Christiansburg, Virginia
  - Ironwood Investigational Site, Lynchburg, Virginia
  - Ironwood Investigational Site, La Crosse, Wisconsin

REFERENCES:
- [Derived] Chey WD, Sayuk GS, Bartolini W, Reasner DS, Fox SM, Bochenek W, Boinpally R, Shea E, Tripp K, Borgstein N. Randomized Trial of 2 Delayed-Release Formulations of Linaclotide in Patients With Irritable Bowel Syndrome With Constipation. Am J Gastroenterol. 2021 Feb 1;116(2):354-361. doi: 10.14309/ajg.0000000000000967. PMID 33065589

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 227 of the 759 participants who signed an informed consent form and entered the Pretreatment Period were not randomized into the study, and were identified as pretreatment failures.
Groups:
- Placebo: Placebo: once daily (QD) for 12 weeks
- Linaclotide IR 290 μg: Linaclotide immediate release (IR) formulation: 290 μg QD for 12 weeks
- Linaclotide DR1 30 μg: Linaclotide delayed release formulation 1 (DR1) 30 μg QD for 12 weeks
- Linaclotide DR1 100 μg: Linaclotide DR1 100 μg QD for 12 weeks
- Linaclotide DR1 300 μg: Linaclotide DR1 300 μg QD for 12 weeks
- Linaclotide DR2 30 μg: Linaclotide delayed release formulation 2 (DR2) 30 μg QD for 12 weeks
- Linaclotide DR2 100 μg: Linaclotide DR2 100 μg QD for 12 weeks
- Linaclotide DR2 300 μg: Linaclotide DR2 300 μg QD for 12 weeks
Period: Overall Study
Arm/Group | Placebo | Linaclotide IR 290 μg | Linaclotide DR1 30 μg | Linaclotide DR1 100 μg | Linaclotide DR1 300 μg | Linaclotide DR2 30 μg | Linaclotide DR2 100 μg | Linaclotide DR2 300 μg
Started (Randomized) | 66 | 66 | 67 | 67 | 67 | 67 | 66 | 66
Completed | 58 | 54 | 58 | 53 | 55 | 53 | 60 | 57
Not Completed | 8 | 12 | 9 | 14 | 12 | 14 | 6 | 9
Not completed — Adverse Event | 0 | 4 | 1 | 5 | 3 | 0 | 1 | 0
Not completed — Protocol Violation | 1 | 0 | 1 | 0 | 0 | 2 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 3 | 1 | 3 | 5 | 4 | 1 | 2
Not completed — Lost to Follow-up | 3 | 5 | 3 | 3 | 2 | 5 | 1 | 4
Not completed — Lack of Efficacy | 1 | 0 | 3 | 2 | 2 | 3 | 3 | 3
Not completed — Other Not Specified | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Linaclotide IR 290 μg: Linaclotide IR formulation: 290 μg QD for 12 weeks
- Linaclotide DR1 30 μg: Linaclotide DR1 30 μg QD for 12 weeks
- Linaclotide DR2 30 μg: Linaclotide DR2 30 μg QD for 12 weeks
- Total: Total of all reporting groups
Arm/Group | Placebo | Linaclotide IR 290 μg | Linaclotide DR1 30 μg | Linaclotide DR1 100 μg | Linaclotide DR1 300 μg | Linaclotide DR2 30 μg | Linaclotide DR2 100 μg | Linaclotide DR2 300 μg | Total
Number analyzed (Participants) | 66 | 66 | 67 | 67 | 67 | 67 | 66 | 66 | 532
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.4 (14.7) | 44.1 (14.4) | 44.8 (14.9) | 44.7 (13.7) | 46.5 (12.7) | 42.3 (12.6) | 47.9 (12.8) | 45.2 (14.4) | 45.1 (13.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53 | 53 | 59 | 59 | 55 | 50 | 52 | 62 | 443
  Male | 13 | 13 | 8 | 8 | 12 | 17 | 14 | 4 | 89
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 14 | 16 | 17 | 16 | 18 | 15 | 21 | 127
  Not Hispanic or Latino | 56 | 52 | 51 | 50 | 51 | 49 | 51 | 45 | 405
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 38 | 43 | 45 | 47 | 41 | 42 | 40 | 48 | 344
  Non-Caucasian | 28 | 23 | 22 | 20 | 26 | 25 | 26 | 18 | 188
  Black/African American | 25 | 11 | 18 | 17 | 19 | 19 | 22 | 14 | 145
  Asian | 2 | 10 | 3 | 2 | 7 | 6 | 2 | 3 | 35
  Other, Not Specified | 1 | 2 | 1 | 1 | 0 | 0 | 2 | 1 | 8
Abdominal Pain [Mean (Standard Deviation); unit: units on a scale] — Based on 11-point numerical rating scale assessing symptom "at its worst in past 24 hours." 0=No symptom; 10=Worst possible.
  units on a scale | 6.41 (1.85) | 6.18 (1.77) | 6.20 (1.59) | 6.18 (1.67) | 6.38 (1.82) | 6.07 (1.68) | 6.48 (1.53) | 6.09 (1.68) | 6.25 (1.69)
Complete Spontaneous Bowel Movement (CBSM) Weekly Rate [Mean (Standard Deviation); unit: CBSM/week] | 0.29 (0.56) | 0.34 (0.61) | 0.35 (0.56) | 0.22 (0.46) | 0.27 (0.54) | 0.35 (0.62) | 0.31 (0.61) | 0.33 (0.56) | 0.31 (0.57)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Weekly Abdominal Pain Score Over the 12-Week Treatment Period: DR1 or IR vs. Placebo
Description: Abdominal pain assessment was based on an 11-point numerical rating scale (0=No symptom; 10=Worst possible) assessing the symptom "at its worst in past 24 hours." A participant's weekly abdominal pain score is the average of the nonmissing abdominal pain scores reported by the participant during each week.
Time Frame: Baseline, up to Week 12
Population: Intent to Treat Population: all randomized participants who received at least one dose of study drug (evaluated according to assigned treatment).
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Groups:
- Placebo: Placebo: QD for 12 weeks
Arm/Group | Placebo | Linaclotide IR 290 μg | Linaclotide DR1 30 μg | Linaclotide DR1 100 μg | Linaclotide DR1 300 μg
Number analyzed (Participants) | 66 | 66 | 67 | 67 | 67
score on a scale | -1.370 (0.241) | -1.938 (0.241) | -1.667 (0.234) | -1.656 (0.240) | -2.140 (0.236)
Statistical Analysis 1: Comparison: Placebo vs Linaclotide IR 290 μg; Test type: Superiority; p = 0.0839, mixed model repeated measures (MMRM); LS Mean Difference (Lin-Placebo) = -0.569, 95% CI 2-sided [-1.214 to 0.076]
Statistical Analysis 2: Comparison: Placebo vs Linaclotide DR1 30 μg; Test type: Superiority; p = 0.3661, MMRM; LS Mean Difference (Lin-Placebo) = -0.297, 95% CI 2-sided [-0.942 to 0.348]
Statistical Analysis 3: Comparison: Placebo vs Linaclotide DR1 100 μg; Test type: Superiority; p = 0.3869, MMRM; LS Mean Difference (Lin-Placebo) = -0.286, 95% CI 2-sided [-0.936 to 0.363]
Statistical Analysis 4: Comparison: Placebo vs Linaclotide DR1 300 μg; Test type: Superiority; p = 0.0199, MMRM; LS Mean Difference (Lin-Placebo) = -0.771, 95% CI 2-sided [-1.419 to -0.123]
Statistical Analysis 5: Comparison: Placebo vs Linaclotide DR1 30 μg vs Linaclotide DR1 100 μg vs Linaclotide DR1 300 μg; Test type: Superiority; p = 0.0276, Trend Test — Trend test performed using linear contrast statement for each DR formulation with placebo

2. Primary Outcome: Change From Baseline in Weekly Abdominal Pain Score Over the 12-Week Treatment Period: DR2 or IR vs. Placebo
Description: as for outcome 1
Time Frame: Baseline, up to Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Linaclotide IR 290 μg | Linaclotide DR2 30 μg | Linaclotide DR2 100 μg | Linaclotide DR2 300 μg
Number analyzed (Participants) | 66 | 66 | 67 | 66 | 66
score on a scale | -1.370 (0.241) | -1.938 (0.241) | -1.825 (0.238) | -1.669 (0.235) | -1.628 (0.239)
Statistical Analysis 1: Comparison: Placebo vs Linaclotide IR 290 μg; Test type: Superiority; p = 0.0839, MMRM; LS Mean Difference (Lin-Placebo) = -0.569, 95% CI 2-sided [-1.214 to 0.076]
Statistical Analysis 2: Comparison: Placebo vs Linaclotide DR2 30 μg; Test type: Superiority; p = 0.1669, MMRM; LS Mean Difference (Lin-Placebo) = -0.455, 95% CI 2-sided [-1.102 to 0.191]
Statistical Analysis 3: Comparison: Placebo vs Linaclotide DR2 100 μg; Test type: Superiority; p = 0.3637, MMRM; LS Mean Difference (Lin-Placebo) = -0.299, 95% CI 2-sided [-0.947 to 0.348]
Statistical Analysis 4: Comparison: Placebo vs Linaclotide DR2 300 μg; Test type: Superiority; p = 0.4333, MMRM; LS Mean Difference (Lin-Placebo) = -0.258, 95% CI 2-sided [-0.905 to 0.389]
Statistical Analysis 5: Comparison: Placebo vs Linaclotide DR2 30 μg vs Linaclotide DR2 100 μg vs Linaclotide DR2 300 μg; Test type: Superiority; p = 0.5528, Trend Test — Trend test performed using linear contrast statement for each DR formulation with placebo

3. Primary Outcome: Change From Baseline in Weekly CSBM Frequency Rate Over the 12-Week Treatment Period: DR1 or IR vs. Placebo
Description: A participant's weekly CSBM frequency rate is the CSBM rate (CSBMs/week) calculated over that week.
Time Frame: Baseline, up to Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: CSBMs/week
Arm/Group | Placebo | Linaclotide IR 290 μg | Linaclotide DR1 30 μg | Linaclotide DR1 100 μg | Linaclotide DR1 300 μg
Number analyzed (Participants) | 66 | 66 | 67 | 67 | 67
CSBMs/week | 1.115 (0.285) | 2.107 (0.286) | 1.163 (0.278) | 1.414 (0.283) | 1.776 (0.279)
Statistical Analysis 1: Comparison: Placebo vs Linaclotide IR 290 μg; Test type: Superiority; p = 0.0110, MMRM; LS Mean Difference (Lin-Placebo) = 0.992, 95% CI 2-sided [0.228 to 1.756]
Statistical Analysis 2: Comparison: Placebo vs Linaclotide DR1 30 μg; Test type: Superiority; p = 0.9013, MMRM; LS Mean Difference (Lin-Placebo) = 0.048, 95% CI 2-sided [-0.716 to 0.812]
Statistical Analysis 3: Comparison: Linaclotide DR1 100 μg; Test type: Superiority; p = 0.4447, MMRM; LS Mean Difference (Lin-Placebo) = 0.299, 95% CI 2-sided [-0.469 to 1.067]
Statistical Analysis 4: Comparison: Placebo vs Linaclotide DR1 300 μg; Test type: Superiority; p = 0.0904, MMRM; LS Mean Difference (Lin-Placebo) = 0.662, 95% CI 2-sided [-0.104 to 1.428]
Statistical Analysis 5: Comparison: Placebo vs Linaclotide DR1 30 μg vs Linaclotide DR1 100 μg vs Linaclotide DR1 300 μg; Test type: Superiority; p = 0.0700, Trend Test — Trend test performed using linear contrast statement for each DR formulation with placebo

4. Primary Outcome: Change From Baseline in Weekly CSBM Frequency Rate Over the 12-Week Treatment Period: DR2 or IR vs. Placebo
Description: A participant's weekly CSBM frequency rate is the CSBM rate (CSBMs/week) calculated over that week.
Time Frame: Baseline, up to Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: CSBMs/week
Arm/Group | Placebo | Linaclotide IR 290 μg | Linaclotide DR2 30 μg | Linaclotide DR2 100 μg | Linaclotide DR2 300 μg
Number analyzed (Participants) | 66 | 66 | 67 | 66 | 66
CSBMs/week | 1.115 (0.285) | 2.107 (0.286) | 1.275 (0.282) | 1.019 (0.278) | 0.869 (0.282)
Statistical Analysis 1: Comparison: Placebo vs Linaclotide IR 290 μg; Test type: Superiority; p = 0.0110, MMRM; LS Mean Difference (Lin-Placebo) = 0.992, 95% CI 2-sided [0.228 to 1.756]
Statistical Analysis 2: Comparison: Placebo vs Linaclotide DR2 30 μg; Test type: Superiority; p = 0.6801, MMRM; LS Mean Difference (Lin-Placebo) = 0.161, 95% CI 2-sided [-0.604 to 0.925]
Statistical Analysis 3: Comparison: Placebo vs Linaclotide DR2 100 μg; Test type: Superiority; p = 0.8069, MMRM; LS Mean Difference (Lin-Placebo) = -0.095, 95% CI 2-sided [-0.861 to 0.670]
Statistical Analysis 4: Comparison: Placebo vs Linaclotide DR2 300 μg; Test type: Superiority; p = 0.5275, MMRM; LS Mean Difference (Lin-Placebo) = -0.246, 95% CI 2-sided [-1.011 to 0.519]
Statistical Analysis 5: Comparison: Placebo vs Linaclotide DR2 30 μg vs Linaclotide DR2 100 μg vs Linaclotide DR2 300 μg; Test type: Superiority; p = 0.4201, Trend Test — Trend test performed using linear contrast statement for each DR formulation with placebo

5. Primary Outcome: Number of 6/12 Week Abdominal Pain and Constipation (APC) +1 Responders Over the 12-Week Treatment Period: DR1 or IR vs. Placebo
Description: A 6/12 Week APC +1 Responder is a participant who meets the Weekly APC +1 Responder criteria for at least 6 out of the 12 weeks of the Treatment Period.
  * Weekly APC +1 Responder: A participant who meets the criteria to be a Weekly Abdominal Pain Responder and a Weekly CSBM +1 Responder.
  * Weekly Abdominal Pain Responder: A participant who has a decrease from baseline of ≥30% in the mean daily worst abdominal pain scores for that week.
  * Weekly CSBM +1 Responder: A participant who has an increase from baseline of ≥1 in the CSBM weekly rate for that week.
  A participant with <4 days of completed eDiary data for that week is not considered a responder for that week.
Time Frame: up to Week 12
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Linaclotide IR 290 μg | Linaclotide DR1 30 μg | Linaclotide DR1 100 μg | Linaclotide DR1 300 μg
Number analyzed (Participants) | 66 | 66 | 67 | 67 | 67
Participants
  Responder | 14 | 21 | 18 | 17 | 26
  Non-Responder | 52 | 45 | 49 | 50 | 41
Statistical Analysis 1: Comparison: Placebo vs Linaclotide IR 290 μg; Test type: Superiority; p = 0.1663, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.71, 95% CI 2-sided [0.79 to 3.70]
Statistical Analysis 2: Comparison: Placebo vs Linaclotide DR1 30 μg; Test type: Superiority; p = 0.4399, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.39, 95% CI 2-sided [0.61 to 3.17]
Statistical Analysis 3: Comparison: Placebo vs Linaclotide DR1 100 μg; Test type: Superiority; p = 0.5540, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.27, 95% CI 2-sided [0.57 to 2.85]
Statistical Analysis 4: Comparison: Placebo vs Linaclotide DR1 300 μg; Test type: Superiority; p = 0.0262, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 2.39, 95% CI 2-sided [1.10 to 5.19]
Statistical Analysis 5: Comparison: Placebo vs Linaclotide DR1 30 μg vs Linaclotide DR1 100 μg vs Linaclotide DR1 300 μg; Test type: Superiority; p = 0.0249, Correlation test — For each DR formulation, the Correlation Test p-values are obtained from the correlation statistic controlling for geographic region

6. Primary Outcome: Number of 6/12 Week Abdominal Pain and Constipation (APC) +1 Responders Over the 12-Week Treatment Period: DR2 or IR vs. Placebo
Description: as for outcome 5
Time Frame: up to Week 12
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Linaclotide IR 290 μg | Linaclotide DR2 30 μg | Linaclotide DR2 100 μg | Linaclotide DR2 300 μg
Number analyzed (Participants) | 66 | 66 | 67 | 66 | 66
Participants
  Responder | 14 | 21 | 16 | 16 | 14
  Non-Responder | 52 | 45 | 51 | 50 | 52
Statistical Analysis 1: Comparison: Placebo vs Linaclotide IR 290 μg; Test type: Superiority; p = 0.1663, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.71, 95% CI 2-sided [0.79 to 3.70]
Statistical Analysis 2: Comparison: Placebo vs Linaclotide DR2 30 μg; Test type: Superiority; p = 0.7710, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.13, 95% CI 2-sided [0.49 to 2.58]
Statistical Analysis 3: Comparison: Placebo vs Linaclotide DR2 100 μg; Test type: Superiority; p = 0.8021, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.11, 95% CI 2-sided [0.48 to 2.58]
Statistical Analysis 4: Comparison: Placebo vs Linaclotide DR2 300 μg; Test type: Superiority; p = 0.8011, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.89, 95% CI 2-sided [0.37 to 2.14]
Statistical Analysis 5: Comparison: Placebo vs Linaclotide DR2 30 μg vs Linaclotide DR2 100 μg vs Linaclotide DR2 300 μg; Test type: Superiority; p = 0.8578, Correlation test — [p-value comment as in outcome 5, analysis 5]

ADVERSE EVENTS:
Time Frame: From the first dose of study drug through Week 12/End-of-Treatment Period Visit (Day 85+3)
Arm/Group | Placebo | Linaclotide IR 290 μg | Linaclotide DR1 30 μg | Linaclotide DR1 100 μg | Linaclotide DR1 300 μg | Linaclotide DR2 30 μg | Linaclotide DR2 100 μg | Linaclotide DR2 300 μg
All-Cause Mortality (participants affected / at risk) | 0/66 | 0/66 | 0/67 | 0/67 | 0/67 | 0/67 | 0/66 | 0/66
Serious Adverse Events (participants affected / at risk) | 1/66 | 1/66 | 0/67 | 0/67 | 0/67 | 0/67 | 0/66 | 0/66
Other Adverse Events (participants affected / at risk) | 1/66 | 10/66 | 4/67 | 9/67 | 8/67 | 0/67 | 1/66 | 2/66
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=66) | Linaclotide IR 290 μg (N=66) | Linaclotide DR1 30 μg (N=67) | Linaclotide DR1 100 μg (N=67) | Linaclotide DR1 300 μg (N=67) | Linaclotide DR2 30 μg (N=67) | Linaclotide DR2 100 μg (N=66) | Linaclotide DR2 300 μg (N=66)
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=66) | Linaclotide IR 290 μg (N=66) | Linaclotide DR1 30 μg (N=67) | Linaclotide DR1 100 μg (N=67) | Linaclotide DR1 300 μg (N=67) | Linaclotide DR2 30 μg (N=67) | Linaclotide DR2 100 μg (N=66) | Linaclotide DR2 300 μg (N=66)
Diarrhea (Gastrointestinal disorders) | 1 | 9 | 2 | 5 | 7 | 0 | 1 | 2
Headache (Nervous system disorders) | 0 | 1 | 2 | 4 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI may publish or disclose the results of the study 24 months after final data lock provided that sponsor can review the publication prior to public release, sponsor can request removal of confidential information of sponsor (not including results of trial), and sponsor can request a publication delay in order to protect potentially patentable information. Furthermore, if a publication committee is developing an initial publication, PI is to delay disclosure until that publication is published.

DOCUMENTS (2):
  • Statistical Analysis Plan (2016-10-04): https://cdn.clinicaltrials.gov/large-docs/06/NCT02559206/SAP_000.pdf
  • Study Protocol (2015-10-09): https://cdn.clinicaltrials.gov/large-docs/06/NCT02559206/Prot_001.pdf